CLINICAL TRIAL: NCT01545830
Title: Randomized, Controlled Trial of Vitamin D Replenishment in Metabolic Syndrome
Brief Title: Metabolic Syndrome and Insulin Resistance at Allina
Acronym: MISURA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Jeffery Dusek, Senior Consultant, Allina Center for Healthcare Research and Innovation, Allina Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPA ID 3607
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Insulin resistance; Vitamin D deficiency
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Dose (Active Comparator): Intervention: 600 IUs of cholecalciferol taken by mouth daily.
  Interventions: Dietary Supplement: vitamin D3 (cholecalciferol)
- High Dose D (Experimental): Intervention: 6,000 IUs of cholecalciferol taken by mouth daily.
  Interventions: Dietary Supplement: vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: vitamin D3 (cholecalciferol) — Active intervention: 6,000 IUs taken by mouth daily for 6 months Active Comparator: 600 IUs taken by mouth daily for 6 months
  Other Names: D-Drops

SUMMARY:
Vitamin D deficiency is widespread and appears to represent one easily and inexpensively modifiable risk factor for diabetes and cardiovascular disease. More than 40 years of data link hypovitaminosis D to metabolic syndrome, insulin resistance, hyperglycemia, type 2 diabetes and increased cardiovascular risk.

Screening for vitamin D deficiency followed by supplementation in appropriate individuals could be among the simplest and most cost-effective measures for reducing metabolic syndrome and insulin resistance in the general population.

This study will test the hypothesis that increasing vitamin D status in vitamin D deficient individuals with metabolic syndrome will:

1. reduce multiple serum cardiometabolic risk factors for both diabetes and cardiovascular disease,
2. stabilize or reverse the stage of pre-diabetes,
3. improve quality of life, and,
4. improve the ability to make health-related behavioral changes.

DETAILED DESCRIPTION:
Longitudinal observational studies suggest a significant inverse association between vitamin D status and both incident and prevalent metabolic syndrome/type II diabetes. Results from small underpowered trials and post-hoc analyses of data from larger trials designed for bone-specific outcomes suggest that vitamin D may slow the progression to diabetes in adults with glucose intolerance. However, at this time, no randomized trials of sufficient size exist to assess effectiveness.

Importantly, in the investigators' own study of over 10,000 Allina employees, the investigators found that 6% of these employees had levels less than 10 ng/mL, 30% less than 20 ng/ml and 60% less than 30 ng/ml. Recently, the Intermountain Heart Collaborative Study Group reviewed 41,504 patient records with at least one measured vitamin D level. Surprisingly, both the Intermountain and the Allina Employee study demonstrate vitamin D deficiency (≤30 ng/ml) in more than 60% of people tested with only minor differences by gender or age (Plotnikoff GA, Finch M, Dusek JA. Impact of Vitamin D Deficiency on the Productivity of a Health Care Workforce. J Occup Environ Med (in press)).

Furthermore, the Intermountain group demonstrated that vitamin D levels less than 30 ng/ml, compared to levels greater than 30 ng/ml, were associated with highly significant (p <0.0001) increases in the prevalence of diabetes, hypertension, hyperlipidemia, and peripheral vascular disease. Also, those without risk factors but with severe deficiency had an increased likelihood of developing diabetes, hypertension, and hyperlipidemia. The vitamin D levels were also highly associated with coronary artery disease, myocardial infarction, heart failure, and stroke (all p <0.0001), as well as with incident death, heart failure, coronary artery disease/myocardial infarction (all p <0.0001), stroke (p = 0.003), and their composite (p <0.0001).

Numerous prevention efforts are underway to minimize the predicted economic and human burdens from these increasingly common diseases. However, few, if any, prospective clinical trials are underway with vitamin D interventions. This trial is specifically designed to prospectively test the impact of vitamin D replenishment on both metabolic syndrome and insulin resistance.

The 2011 Endocrine Society guidelines assert that vitamin D intakes above the current recommendations may be associated with better health outcomes. However, there is no consensus on the optimal 25(OH)D concentration necessary to minimize metabolic syndrome, insulin resistance and progression to diabetes. This trial is designed to prospectively identify optimal serum levels for reduction of cardiometabolic risk factors.

ELIGIBILITY:
Please Note: All participants must be an employee of Allina Health or the spouse of an Allina employee.

Inclusion Criteria:

* Vitamin D deficiency, defined as 25-OH vitamin D ≤ 25 ng/ml
* Metabolic syndrome as defined by more than three or more of the following:

Elevated waist circumference

* Men - Equal to or greater than 40 inches
* Women - Equal to or greater than 35 inches
* Elevated serum triglycerides (≥150 mg/dL)
* Men - Less than 40 mg/dL
* Women - Less than 50 mg/dL
* Elevated blood pressure (≥130/85 or use of medication for hypertension)
* Elevated fasting glucose (≥100 mg/dL or use of medication for hyperglycemia)

Exclusion Criteria:

* Known cardiovascular disease defined as current or prior coronary heart disease, stroke/transient ischemic attack, heart failure, or peripheral vascular disease.
* During the study, addition of any medications known to change outcome measures including medications or supplements for hyperlipidemia, hypertension, weight loss, diabetes.
* Current Vitamin D supplementation beyond that found in a multivitamin (400 IU)
* Current calcium supplementation greater than 600 mg
* Untreated blood pressure greater than 159/99 at baseline
* Treated blood pressure greater than 150/90 at baseline
* Any condition which could limit the ability to complete and comply with 6-month study
* Unwillingness or inability to comply with study requirements
* Known allergy to coconut or coconut oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
insulin resistance score by NMR lipid fractionation | 6 months
  additional insulin resistance measure
Reynolds Risk Score | 6 months
  The Reynolds Risk Score is designed to predict one's risk of having a future heart attack, stroke, or other major heart disease in the next 10 years. In addition to your age, blood pressure, cholesterol levels and whether you currently smoke, the Reynolds Risk Score uses information from two other risk factors, a blood test called hsCRP (a measure of inflammation) and whether or not either of your parents had a heart attack before they reached age 60 (a measure of genetic risk).
Pre-diabetes stage | 6 months
  The pre-diabetes stage, a marker of progression toward type 2 diabetes mellitus, is a calculated score based upon results of fasting adiponectin, insulin and proinsulin.

SECONDARY OUTCOMES:
25-OH-vitamin D | 6 months
  25-OH-vitamin D is the best measure of vitamin D status.
fasting lipid profile | 6 months
adiposity markers | 6 months
  Adiponectin: This adipocyte-derived protein increases hepatic and peripheral insulin sensitivity, moderates fat tissue growth, decreases lipid and glucose production in the liver and suppresses vascular inflammation. This measure declines as insulin resistance increases.
  Leptin: This adipocyte-derived hormone plays a key role in regulating neuroendocrine and immune function, appetite, metabolic rate and body weight. Many overweight individuals have elevated levels and leptin resistance.
TNF-alpha | 6 months
  Inflammatory markers: TNF-alpha, IL-6, IL-8. These inflammatory mediators are central to the pathophysiology of obesity and its systemic effects
weight | 6 months
blood pressure | 6 months
PROMIS-29 | 6 months
  PROMIS is a questionnaire data bank developed and made available by the National Institutes of Health for research purposes. It is used to measure the core domains of physical functioning, fatigue, pain, depression, anxiety, and social role participation.
Perceived Stress Scale (PSS) | 6 months
  The PSS is brief, validated and widely used psychological instrument for assessing a participant's perception of stress. The PSS-4 consists of 4 questions to measure the degree to which situations in the participant's life are perceived as stressful including questions related to perceived unpredictability and lack of control.
WPAI | 6 months
  This 6 item, validated instrument measures work and general activity impairment due to health problems. It uses a seven day recall and has been adapted for use in populations with differing health problems.
PROMIS-GH | 6 months
  PROMIS is a questionnaire data bank developed and made available by the National Institutes of Health for research purposes. The PROMIS-GH consists of 10 items, representing multiple domains and can be scored into a Global Physical Health component and a Global Mental Health component
International Physical Activity Questionnaire (IPAQ) | 6 months
  The International Physical Activity Questionnaire (IPAQ) short form (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaire is to provide a common instrument that can be used to obtain internationally comparable data on health related physical activity. The development of this international measure for physical activity commenced in Geneva in 1998 and was followed by extensive reliability and validity testing undertaken in 12 countries (14 sites) across 6 continents during 2000.
IL-6 | 6 months
  Inflammatory mediators, including IL-6, are central to the pathophysiology of obesity and its systemic effects.
IL-8 | 6 months
  Inflammatory mediators, inlcuding IL-8, are central to the pathophysiology of obesity and its systemic effects.
HS-CRP | 6 months
  Elevated HS-CRP predicts the development of type II diabetes and is a crucial factor in calculating the Reynolds Risk Score.
Lp-PLA2 (PLAC) | 6 months
  This is an enzyme produced by inflammatory cells that hydrolyzes oxidized phospholipids in HDL and catalyzes the degradation of PAF, platelet activating factor. Levels are positively correlated with increased risk of developing coronary artery disease and stroke.
PAI-1 | 6 months
  This is the primary inhibitor of plasminogen activation. Elevated levels predispose to clot formation by inhibiting fibrinolytic activity.
Fibrinogen | 6 months
  Fibrinogen is also known as coagulation Factor I. Elevated levels are associated with cardiovascular disease. This is an acute-phase protein that is elevated in any form of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Plotnikoff, MD, Principal Investigator — Allina Health; Jeffery Dusek, PhD, Study Director — Allina Health; Shaina Biron, Study Director — Allina Health
Locations (1):
- Allina Health, Minneapolis, Minnesota, United States